CLINICAL TRIAL: NCT03986398
Title: Nosocomial Infections During Total Prostatic Cystectomies (TPC) With Replacement Enterocystoplasty: Prophylactic Role of Urell®, Cranberry Fruit Juice Extract (Vaccicium Macrocarpon)
Acronym: Cranberry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In the perioperative setting of radical cystectomy-bladder replacement no improvement of UTI was noticed in 10 patients who took Urell following the protocol
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018045
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prophylactic efficacy of Urell® (Experimental): Prophylactic efficacy of Urell® on urinary tract infections in patients with bladder cancer and total prostatic cystectomy with replacement enterocystoplasty
  Interventions: Other: Infection prophylaxis

INTERVENTIONS:
Other: Infection prophylaxis — Infection prophylaxis with Urell®, cranberry fruit juice extract (vaccinium macrocarpon)

SUMMARY:
Total prostatic cystectomy with enterocystoplasty is the most extensive urological surgical procedure and one with the highest complication rate, especially infectious complication. The mortality rate remains substantial (2 to 5%).

Examination of hundreds of TPCs made every year in the Urology Department of Foch Hospital, shows that nosocomial urinary infection is constant, especially when the TPC is followed by the constitution of an ileal bladder replacement.

This is due to the intervention itself and duration of postoperative urinary cathéters (ureteral and bladder). This leads to increase surveillance and antibiotic treatment, given the risks of declared infection in this context.

Detailed analysis of the last 20 TPCs with enterocystoplasty showed the presence of germs in significant numbers, in all cases.

Urell® (also sold under the Trademark Ellura®) contains a cranberry juice extract with a high content of bioactive, soluble Proanthocyanidins (PACs) . The daily dose is 36 mg total PACs measured by the DMAC/A2 method. The PACs prevent uropathogenic E.col bacteria from adhering to uroepithelial cells . Their long term use does not create any resistance of the bacteria.

The excellent prophylactic effet of Urell® had been previously observed in the same Center under different conditions.

Therefore a further demonstration was justified, of the prophylactic efficacy of Urell® in the perioperative setting of total prostato-cystectomy with substitute enterocytoplasty, where the slightest urinary infection, symptomatic or not, prolongs hospitalization and requires antibiotic treatment because of its harmful and sometimes major consequences.

ELIGIBILITY:
Inclusion Criteria:

* patient aged > 18 years old
* patient with bladder cancer and total prostatic cystectomy with replacement enterocystoplasty
* signed informed consent
* patient with healthcare insurance

Exclusion Criteria:

* patient without signed informed consent
* patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Number of infectious events | From study treatment start until 21 days of treatment
  Number of symptomatic and non-symptomatic events

SECONDARY OUTCOMES:
Digestive tolerance | From study treatment start until 21 days of treatment
  Assessment on the date of resumption of transit, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Martine Butreau, Principal Investigator — Urology department
Locations (1):
- Hôpital Foch, Suresnes, France